CLINICAL TRIAL: NCT07392164
Title: Speech-Evoked Auditory Potentials: Multisite Pediatric Evaluation
Acronym: SEFR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Susan Scollie (Other)
Collaborators: Dalhousie University (Other)
Responsible Party: Sponsor-Investigator, Susan Scollie, Professor, Western University, Canada
Organization: Western University, Canada (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 122331
Record Dates: First submitted 2025-12-01; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Hearing Impairment
Keywords: Hearing; Hearing impairment; Hearing aids; Evoked potentials; Pediatrics
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Infants with normal hearing and with hearing loss (Experimental): Infants with clinically confirmed normal hearing and hearing loss. Participants will undergo up to 2 recording sessions of speech-evoked envelope following responses (EFRs) using the newly developed prototype device in both unaided (for normal hearing) and aided conditions (if child has been fit with hearing aids). If applicable, hearing aid settings will be recorded; their device settings will not be altered. Hearing assessment results and acoustic measures will be obtained through chart review with caregiver consent.
  Interventions: Device: A newly developed prototype device for speech-evoked EFR Measurement

INTERVENTIONS:
Device: A newly developed prototype device for speech-evoked EFR Measurement — Speech-evoked envelope following responses (EFRs) are measured using the newly developed clinical prototype to objectively assess auditory responses. Surface electrodes are placed on the head, a non-sense speech stimulus is presented at an average level, and EFRs are recorded for 15-30 minutes while patient sleeps or is at rest.

SUMMARY:
The goal of this study is to evaluate the sensitivity of a newly-developed prototype device in its ability to measure brain responses to speech sounds in an infant population. The main research questions are: 1) Is the prototype sensitive to brain response differences from infants with hearing loss with and without hearing aids? and 2) How do the measured brain responses from infants with hearing loss compare to infants with normal hearing who are the same age? Participants will have their brain responses measured using the prototype in response to average-level non-sense speech sounds across 1 to 2 sessions in a "no-hearing aids" condition. Participants with hearing loss who are already fit with hearing aids will additionally undergo a "with hearing aids" recording condition.

DETAILED DESCRIPTION:
In addition to the listed collaborator sites under the "sponsors and collaborators" section, this study is conducted in collaboration with the National Acoustic Laboratories (NAL), Australia, who serve as an international clinical research site contributing to data collection and scientific expertise in pediatric audiology. The prototype is being provided by Audioscan, Dorchester, ON, Canada.

Additionally, the newly developed clinical prototype device is not a U.S. FDA-regulated device. ClinicalTrials.gov registration is being completed as a prerequisite for Health Canada's investigational testing of medical devices, as outlined in Health Canada's 2007 Notice concerning registration and public disclosure of clinical trial information. The application number for Health Canada's investigational testing authorization is 389562.

ELIGIBILITY:
Inclusion Criteria:

1. Infants (3 to 24 months of age) with normal hearing who have passed their audiological diagnostic evaluation
2. Infants (3 to 24 months of age) identified with hearing loss at their audiological diagnostic evaluation, whose parents have chosen spoken language as their form of communication, and who have been prescribed and fitted with a hearing aid(s).

Exclusion Criteria:

Participants who have abnormal middle ear measure results or occluding ear wax will be excluded.

Ages: 3 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Speech-Evoked Envelope Following Responses (EFRs) Agreement with Hearing Assessment | Outcomes are assessed during the initial recording session (Day 1). When two sessions are required, outcome data collection is completed within 2 weeks of the first session.
  EFR detection rates will be compared to hearing assessment results for the "Infants with normal hearing" and the "Infants with hearing loss" group for the unaided recording condition. Correlation and regression analysis will be used to look at agreement between prototype measures and the child's hearing assessment results.

SECONDARY OUTCOMES:
Speech-evoked Envelope Following Response (EFR) Amplitude in Infants with Hearing Loss | Outcomes are assessed during the initial recording session (Day 1). When two sessions are required, outcome data collection is completed within 2 weeks of the first session.
  EFR amplitudes will be compared between the aided and unaided conditions of the "Infants with hearing loss" group. Repeated measures ANOVA and post-hoc paired t-tests will be used for data analysis.
Speech-Evoked Envelope Following Responses (EFRs) Amplitude Between Normal Hearing and Hearing Loss Infants | Outcomes are assessed during the initial recording session (Day 1). When two sessions are required, outcome data collection is completed within 2 weeks of the first session.
  EFR amplitudes will be compared between the "Infants with normal hearing" and the "Infants with hearing loss" groups. EFR amplitude will also be compared between groups by deriving a normal range of measurement (from normal hearing infants) and characterizing whether measures from infants with hearing loss are or are not within that range. This is a descriptive, not inferential, analysis that is mainly used to aid in interpretation of the nature of the response, so inferential statistics are not proposed.
Speech-evoked Envelope Following Response (EFR) detection rates in Infants with Hearing Loss | Outcomes are assessed during the initial recording session (Day 1). When two sessions are required, outcome data collection is completed within 2 weeks of the first session.
  EFR detection rates will be compared between the aided and unaided conditions of the "Infants with hearing loss" group. Repeated measures ANOVA and post-hoc paired t-tests will be used for data analysis.
Speech-Evoked Envelope Following Responses (EFRs) Detection Rate Between Normal Hearing and Hearing Loss Infants | Outcomes are assessed during the initial recording session (Day 1). When two sessions are required, outcome data collection is completed within 2 weeks of the first session.
  EFR detection rate will be compared between the "Infants with normal hearing" and the "Infants with hearing loss" groups. EFR detection rate will also be compared between groups by deriving a normal range of measurement (from normal hearing infants) and characterizing whether measures from infants with hearing loss are or are not within that range. This is a descriptive, not inferential, analysis that is mainly used to aid in interpretation of the nature of the response, so inferential statistics are not proposed.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Scollie, PhD, Principal Investigator — Western University; David Purcell, PhD, Principal Investigator — Western University
Locations (3):
- National Acoustic Laborartory, Macquarie Park, Sydney, Australia
- Canada (2):
  - Dalhousie University, Halifax, Nova Scotia
  - National Centre for Audiology at Western University, London, Ontario

IPD SHARING:
Plan to Share IPD: Yes
For the reasons of transparency and education, it is strongly encouraged by many medical journals and other authorities to publish the anonymized data from clinical studies for public use. This data is visible to researchers or the general public after the study is over. Researchers may use this data to improve knowledge about brain responses to speech sounds.
  We will publish the following anonymized data from this study: audiogram, middle ear analysis, speech test scores, and auditory evoked potentials. Note that there will be NO personal identifiers in this list.
Supporting Information: SAP, CSR
Time Frame: The de-identified IPD and supporting information will be available beginning immediately after publication, with no end date.
Access Criteria: Access to individual participant data will be restricted to authorized research personnel directly involved in data collection, compilation, and analysis at Western University, Dalhousie University, and the National Acoustics Laboratories. Each site will retain identifiable information locally, including consent forms and master lists, which will not be shared. Only de-identified data will be uploaded to a secure, password-protected SharePoint system hosted by Western University for shared analysis. The industry partner (Audioscan) may receive de-identified technical output only if needed for prototype improvement. No identifiable information will be released externally, and results will be reported in aggregate form only.
URL: https://www.bmj.com/open-data

REFERENCES:
- [Background] Easwar, V., Scollie, S., Lasarev, M., Urichuk, M., Aiken, S.J., Purcell, D.W. (2021). Characteristics of speech-evoked envelope following responses in infancy. Trends in Hearing. Published online doi: 10.1177/23312165211004331
- [Background] Easwar, V., Purcell, D., Aiken, S., Parsa, V., Scollie, S. (2015). Evaluation of speech-evoked envelope following responses as an objective aided outcome measure: Effect of stimulus level, bandwidth, and amplification in adults with hearing loss. Ear and Hearing, Published online doi: 10.1097/AUD.0000000000000188.